CLINICAL TRIAL: NCT06306573
Title: CardioMEMS™ HF System Real-World Evidence Post-Approval Study
Brief Title: CardioMEMS HF System Real-World Evidence Post-Approval Study
Status: Enrolling by invitation | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: CL1019613
Record Dates: First submitted 2023-11-14; First posted 2024-03-12 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Heart Failure NYHA Class II; Heart Failure NYHA Class III
Keywords: CardioMEMS HF System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Primary Cohort: The Primary Cohort will include NYHA Class II heart failure subjects receiving a CardioMEMS PA Sensor implant in the commercial setting.
  Interventions: Device: CardioMEMS HF System
- Full Cohort: The Full Cohort will include both NYHA Class II and Class III heart failure subjects receiving a CardioMEMS PA Sensor implant in the commercial setting.
  Interventions: Device: CardioMEMS HF System

INTERVENTIONS:
Device: CardioMEMS HF System — The CardioMEMS HF System provides pulmonary artery (PA) hemodynamic data to monitor and manage HF subjects. The CardioMEMS HF System measures PA pressure which clinicians use to initiate or modify HF treatment.

SUMMARY:
The purpose of this post-approval study (PAS) is to evaluate the long-term safety and effectiveness of the CardioMEMS™ HF System using real-world evidence (RWE) methods.

DETAILED DESCRIPTION:
Subjects will be identified in Abbott's Merlin.net remote monitoring database. Merlin.net data will be linked to Medicare fee-for-service (FFS) claims data to longitudinally track outcomes. Each subject will be followed for a minimum of 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Subject implanted with a CardioMEMS PA Sensor and enrolled in Merlin.net
* Subject resides in the United States as documented in Merlin.net
* NYHA Class II or Class III as documented in Merlin.net at the time of CardioMEMS implant (only NYHA Class II subjects contribute to the Primary Cohort)
* Subject identified in Merlin.net data can be linked to Medicare FFS claims
* Subject is enrolled in Medicare Part A and B, and not enrolled in Medicare Part C, at implant and for 12 months prior to implant, to establish qualification for CardioMEMS
* Subject ≥18 years of age at time of CardioMEMS implant

Exclusion Criteria:

* Subject received heart transplant or durable mechanical circulatory support device implant (i.e., left/right/bi-ventricular assist device) prior to CardioMEMS implant

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The intended population for this RWE PAS includes Medicare FFS beneficiaries with symptomatic NYHA Class II and III heart failure implanted with a CardioMEMS PA Sensor in the commercial setting.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Two-Year Survival in the Primary Cohort (NYHA Class II subjects) | 2 years
  Evaluate survival for the Primary Cohort compared to a pre-specified performance goal of 71.7% survival at 2 years.

SECONDARY OUTCOMES:
Two-Year Survival in the Full Cohort (NYHA Class II and Class III subjects) | 2 years
  Evaluate survival for the Full Cohort compared to a pre-specified performance goal of 69.6% survival at 2 years.

OTHER OUTCOMES:
3-Year Survival | 3 years
  Evaluate survival for the Primary and Full Cohorts at 3 years
HF Hospitalization Rate | 3 years
  Evaluate HF hospitalization rates in the Primary and Full Cohorts at 3 years
Pulmonary Artery (PA) Pressures Measured by the CardioMEMS PA Sensor | 3 years
  Systolic, diastolic, and mean PA pressures submitted to Merlin.net from the CardioMEMS PA sensor will be evaluated at fixed timepoints every 6 months (e.g., baseline, 6 months, 12 months, etc) in the Primary and Full Cohorts.
Subject Compliance Rates with Weekly Pulmonary Artery (PA) Pressure Uploads | 3 years
  Subject compliance rates with weekly PA pressure uploads will be evaluated in the Primary and Full Cohorts from 0 to 3 years. The compliance rate will be calculated for each subject as the number weeks with at least 1 PA pressure upload to Merlin.net divided by the total number of weeks of follow-up.
Number of Subjects with Heart Failure (HF) Prescription Medication Fills | 3 years
  The number of patients with prescription claims for HF medications of interest will be reported from 0 - 3 years in the Full Cohort. Data will be reported as the number of subjects who have at least 1 prescription filled for each of the following drug classes during each 6-month interval of follow-up: angiotensin-converting enzyme inhibitor, angiotensin receptor blocker, angiotensin receptor-neprilysin inhibitor, beta blocker, mineralocorticoid receptor antagonist, diuretics, hydralazine, nitrates, and sodium-glucose cotransport-2 inhibitor.
Proportion of Subjects with Heart Failure (HF) Prescription Medication Fills | 3 years
  The proportion of patients with prescription claims for HF medications of interest will be reported from 0 - 3 years in the Full Cohort. Data will be reported as the proportion of subjects who have at least 1 prescription filled for each of the following drug classes during each 6-month interval of follow-up: angiotensin-converting enzyme inhibitor, angiotensin receptor blocker, angiotensin receptor-neprilysin inhibitor, beta blocker, mineralocorticoid receptor antagonist, diuretics, hydralazine, nitrates, and sodium-glucose cotransport-2 inhibitor.

CONTACTS AND LOCATIONS:
Locations (1):
- Abbott Medical, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No